CLINICAL TRIAL: NCT01474642
Title: A Randomized Phase II Trial of Capecitabine Plus Cisplatin (XP) Versus Capecitabine Plus Genexol (XG) as a First-line Treatment for Advanced or Recurrent Esophageal Squamous Cell Carcinoma
Brief Title: Phase II Trial of XP Versus XG in Advanced Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-09-10
Record Dates: First submitted 2011-11-10; First posted 2011-11-18 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Advanced or Recurrent Esophageal Squamous Cell Carcinoma
Keywords: Advanced or recurrent esophageal squamous cell carcinoma; Randomizes phase II trial; Capecitabine; Cisplatin; Genexol
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capecitabine/Cisplatin(XP) (Active Comparator): Capecitabine AND Cisplatin
  Interventions: Drug: Capecitabine/Cisplatin(XP)
- Capecitabine/Paditaxel(XG) (Active Comparator): Capecitabine + Paditaxel(genexol)
  Interventions: Drug: Capecitabine/Paditaxel(XG)

INTERVENTIONS:
Drug: Capecitabine/Cisplatin(XP) — Capecitabine/Cisplatin(XP) D1-D14 Capecitabine 2000mg/m2 D#2 PO D1 Cisplatin 75mg/m2 iv q 3 weeks
  Arms: Capecitabine/Cisplatin(XP)
Drug: Capecitabine/Paditaxel(XG) — Capecitabine/Paditaxel(XG) D1-D14 Capecitabine 2000mg/m2 D#2 PO D1,D8 Paditaxel(genexol) 80mg/m2 iv q 3 weeks
  Arms: Capecitabine/Paditaxel(XG)

SUMMARY:
Until today, the 5-FU/cisplatin combination is the reference regimen with 30-45% response rates, which is most commonly used to treat patients with metastatic, recurrent or locally advanced, unresectable squamous cell carcinoma of the esophagus. Because the classical dose schedule of this two-drug combination is cisplatin 100 mg/m2 day 1 and 5-FU 1000 mg/m2/day continuous infusion for 96-120 hr, prolonged administration time and mucosal toxicity are inconvenient to the patients with the aim of palliation. Capecitabine, which is oral prodrug of 5-FU and mimic continuously-infused 5-FU, is being investigated in phase I, II and III trials for the treatment of gastric, gastroesophageal, and esophageal cancers, primarily in the first-line metastatic setting but also in the adjuvant setting. In the investigators experience, capecitabine plus cisplatin combination (XP) as a first-line treatment for 45 patients with advanced or recurrent esophageal squamous cell carcinoma demonstrated a promising anti-tumor activity with 57% of response rate and showed tolerable toxicity with convenience.

Paclitaxel has been also investigated as monotherapy and in combination with cisplatin in patients with advanced esophageal cancer. A Dutch phase II study demonstrated that paclitaxel combination with carboplatin had shown an encouraging confirmed response rate of 59% with 51 patients with resectable esophageal cancer in neoadjuvant setting. Another Dutch phase II study showed 43% of response rate including 4% of CR with 8 months of response duration when paclitaxel plus cisplatin administration was given for patients with metastatic esophageal cancer. Although recently first-line palliative chemotherapy regimen in esophageal cancer has been investigated, many trials have failed to show superiority to 5-FU/cisplatin combination. Since the investigators considered that XP or XG (genexol) is more effective and convenient chemotherapy regimen than 5-FU/cisplatin, this randomized phase II study was planned to compare XP with XG in terms of efficacy and tolerability.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed metastatic, or recurrent esophageal squamous cell carcinoma
* Age > 18 years
* ECOG performance status 0 - 2
* At least one measurable lesion(s) by RECIST criteria
* Life expectancy ≥ 3 months
* No prior palliative chemotherapy
* Patients may have received prior adjuvant chemotherapy with 5-FU with cisplatin as long as it has been 6months since completion of regimen.
* Adequate bone marrow function (≥ ANC 1,500/ul, ≥ platelet 100,000/ul, ≥ Hb 9.0 g/dl)
* Adequate renal function (≤ serum creatinine 1.5 mg/dl or CCr ≥ 50 ml/min)
* Adequate liver function (≤ serum bilirubin 1.5 mg/dl, ≤ AST/ALT x 3 UNL)
* Written informed consent

Exclusion Criteria:

* Other tumor type than squamous cell carcinoma
* CNS metastasis
* Contraindication to any drug contained in the chemotherapy regimen
* Previous adjuvant treatment with 5-FU, cisplstin, capecitabine or paclitaxel finished less than 1 year6 months
* Evidence of serious gastrointestinal bleeding
* History of another malignancy within the last five years except cured
* basal cell carcinoma of skin and cured carcinoma in-situ of uterine cervix
* Clinically significant cardiac disease
* Serious pulmonary conditions/illness
* Serious metabolic disease such as severe non-compensated diabetes mellitus
* History of significant neurologic or psychiatric disorders
* Serious uncontrolled intercurrent infections, or other serious uncontrolled concomitant disease
* Positive serology for the HIV
* Pregnancy, breast feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-09; Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
response rate | 12 months

SECONDARY OUTCOMES:
progression free survival | 12 months
quality of life | 12 months
Number of Adverse Event | 12 months
overall survival | 12 months
predictive marker | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, M.D., Ph.D., Principal Investigator — Samsung Medical Center, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea